CLINICAL TRIAL: NCT06717178
Title: Correlation of the Cancer and Aging Research Group (CARG) Chemotherapy Toxicity Risk Scores and Unplanned Hospitalizations in Older Cancer Patients--A Multi-center Prospective Cohort Study
Brief Title: Cancer and Aging Research Group (CARG) Chemotherapy Toxicity Risk Scores in Older Adults With Cancer in China
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Lirong Yang, Pharmacist, RenJi Hospital
Other Study IDs: LY2024-267-B
Record Dates: First submitted 2024-12-01; First posted 2024-12-04 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Cancer-related Problem/Condition
Keywords: Cancer; Toxicity; Geriatric
MeSH Terms: conditions — Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Chemotherapy — Admission to the hospital for a new chemotherapy regimen (initial or change)

SUMMARY:
The goal of this observational study is to learn about the impact of chemotherapy-related toxicity on older cancer patients in China. The main question it aims to answer is:

Does the Cancer and Aging Research Group (CARG) chemotherapy toxicity risk score predict chemotherapy-related toxicity in Chinese cancer patients over age 70? Participants over age 70 on systemic chemotherapy will answer questions listed in the CARG chemotherapy toxicity risk tool.

DETAILED DESCRIPTION:
Study Background:

There's a high burden of cancer in the geriatric population. Because of factors such as declining organ function, older adults with cancer generally have lower tolerability of chemotherapy than younger patients. In cancer patients aged ≥ 70 years, chemotherapy-related toxic effects were associated with reduced quality of life and/or decreased physical functioning or death after 1 year. Identifying of older patients at high risk of experiencing chemotherapy-related adverse events is one of the key components for developing new prevention and intervention strategies to improve treatment outcomes in older adults with cancer. The CARG toxicity score prediction model and calculator established by the Cancer and Aging Research Group (CARG) in 2011 is widely used in many countries and regions around the world and are recommended by several international guidelines. However, data from older adults with cancer in China are scarce. Prospective studies exploring the correlation between the CARG chemotherapy risk score and unplanned hospitalizations are limited.

Study Objectives:

* To assess the predictive value of the CARG chemotherapy toxicity risk score in older adults with cancer in China
* To explore the correlation between the CARG scores and the unplanned hospitalizations

Study Method:

This is a multi-center prospective cohort study to collect data from cancer patients aged ≥ 70 years from Renji Hospital and Henan Cancer Hospital. Patients will complete the CARG chemotherapy toxicity risk score questionnaires upon initiating a new chemotherapy regimen. The demographics, tumor characteristics (type of cancer and stage), clinical characteristics (e.g. ECOG performance status, NRS-2002 score, and comorbidities), and cancer treatment (e.g. chemotherapy regimen, line of treatment, combined targeted and/or immunotherapy) will be documented for the baseline evaluation. Toxicity, unplanned hospitalization events, and completion of chemotherapy treatment will be assessed for each visit.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 70 years old
* Confirmed diagnosis of solid tumor (any stage)
* ECOG-PS score 0-2 points
* Admission to the hospital for a new chemotherapy regimen (initial or change)
* Patients need to have the ability to read and write, or communicate in Chinese
* The patient must have the ability to give informed consent.

Exclusion Criteria:

* Patients who are on immunotherapy and/or targeted therapy only
* Patients with hematologic malignancy
* Patients with severe infections (sepsis, severe respiratory tract infections, severe urinary tract infections, severe abdominal infections, etc.).
* Patients with severe heart, liver, and kidney dysfunction or failure

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Academic medical centers
Sampling Method: Non-Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Grade 3-5 Chemotherapy-Related Adverse Events as Assessed by CTCAE v4.0 | Each planned admission/unplanned hospitalization until 1 month after completion of chemotherapy or 6 months after the start of chemotherapy
  A grade 3 chemotherapy-related adverse event indicates an event that requires hospitalization. A grade 4 event is life-threatening. A grade 5 event is death.
Number of Participants with Unplanned Hospitalization Events | Each planned admission/unplanned hospitalization until 1 month after completion of chemotherapy or 6 months after the start of chemotherapy
  The unexpected admission to hospital after the initiation of chemotherapy

SECONDARY OUTCOMES:
Number of Participants with Treatment Discontinuation Events | Each planned admission/unplanned hospitalization until 1 month after completion of chemotherapy or 6 months after the start of chemotherapy
  The delivered cycles are fewer than the planned cycles.
Number of Participants with Dose Reduction Events | Each planned admission/unplanned hospitalization until 1 month after completion of chemotherapy or 6 months after the start of chemotherapy
  The dose of at least one chemotherapy drug was reduced by at least 15% compared to standard dose.
Number of Participants with Dose Delay Events | Each planned admission/unplanned hospitalization until 1 month after completion of chemotherapy or 6 months after the start of chemotherapy
  The administration of at least one cytotoxic drug from a chemotherapy regimen was delayed for at least 7 days.
Number of Participants with Dose Missing Events | Each planned admission/unplanned hospitalization until 1 month after completion of chemotherapy or 6 months after the start of chemotherapy
  During the cycle, at least one drug from the chemotherapy regimen is not administered.
Number of Participants with Events of Reduction in Relative Dose Intensity (RDI) | Each planned admission/unplanned hospitalization until 1 month after completion of chemotherapy or 6 months after the start of chemotherapy
  Relative dose intensity (RDI) is the ratio of delivered dose intensity to standard or planned dose intensity. An RDI less than 85% is generally considered to be a clinically significant reduction from standard or planned therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lirong Yang, PharmD, Principal Investigator — Renji Hospital affiliated with Shanghai Jiao Tong University School of Medicine; Xiaoxia Qiu, MS, Principal Investigator — Renji Hospital affiliated with Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Renji Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized individual participant data including clinical characteristics and outcomes will be made available to other researchers on reasonable request.